CLINICAL TRIAL: NCT05082363
Title: The Expression Profile of New Complement Components in Childhood Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Khalifa, principle investigator, Assiut University
Other Study IDs: LNC4D
Record Dates: First submitted 2021-10-07; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- systemic lupus wth renal affection: pt diagnosed with lupus nephritis
  Interventions: Combination Product: C4d evaluation in lupus nephritis in serum and renal tissue
- systemic lupus without renal affection: pt diagnosed as systemic lupus without renal affection
  Interventions: Combination Product: C4d evaluation in lupus nephritis in serum and renal tissue

INTERVENTIONS:
Combination Product: C4d evaluation in lupus nephritis in serum and renal tissue — C4d plasma levels were analyzed by a unique assay specifically detecting C4d arising from complement activation and C4 plasma levels were quantified with competitive ELISA. SLE patients in activitity with and without lupus nephritis In patient with lupus nephritis we will evaluate the C4d after developing remission in the form of reduction of proteinurea less than .5g/g measured as PCR as complete response and less than50% reduction in proteinurea in partial response according to KIDGO guide line Percutaneous renal biopsies were performed in SLE and non-SLE patients under ultrasonographic guidance. 10% formalin-fixed tissue was embedded in paraffin. Four μm-thick sections were stained with hematoxylin and eosin (H&E), periodic acid-Schiff (PAS), periodic acid methenamine silver (PAM), masson-trichrome and polyclonal rabbit anti-human C4d antibody, Renal biopsy specimens of SLE patients were assessed using the most recent modification of the World Health Organization (WHO)

SUMMARY:
The aim of this study was to evaluate whether C4d is a better biomarker and examine whether C4d plasma levels correlate with treatment response and C4d kidney deposition in systemic lupus erythematosus (SLE) with lupus nephritis (LN).

DETAILED DESCRIPTION:
Evaluation of C4d in lupus nephritis in children C4d level difference in children with systemic lupus with and without renal affection C4d level in lupus nephritis at activity and after remission Detection of C4d deposition in renal tissue relation to disease activity

ELIGIBILITY:
Inclusion Criteria:

* This will include children and adolescents who fulfill the 2012 Systemic Lupus International Collaborating Clinics (SLICC)(10) classification criteria of SLE.

  * Inclusion Criteria:

    * Age younger than 18 years.
    * Active SLE with and without renal affection
    * Patients with biopsy proven LN according to ISN/RPS classification criteria of Lupus nephritis.

Exclusion Criteria:

* -Patients in remission.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Age younger than 18 years.
  * Active SLE with and without renal affection
  * Patients with biopsy proven LN according to ISN/RPS classification criteria of Lupus nephritis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of C4d in lupus nephritis in children | 2 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin M, Trattner R, Nilsson SC, Bjork A, Zickert A, Blom AM, Gunnarsson I. Plasma C4d Correlates With C4d Deposition in Kidneys and With Treatment Response in Lupus Nephritis Patients. Front Immunol. 2020 Oct 2;11:582737. doi: 10.3389/fimmu.2020.582737. eCollection 2020. PMID 33133102
- [Background] Bennett M, Brunner HI. Biomarkers and updates on pediatrics lupus nephritis. Rheum Dis Clin North Am. 2013 Nov;39(4):833-53. doi: 10.1016/j.rdc.2013.05.001. Epub 2013 Jul 16. PMID 24182857
- [Background] Kim MK, Maeng YI, Lee SJ, Lee IH, Bae J, Kang YN, Park BT, Park KK. Pathogenesis and significance of glomerular C4d deposition in lupus nephritis: activation of classical and lectin pathways. Int J Clin Exp Pathol. 2013 Sep 15;6(10):2157-67. eCollection 2013. PMID 24133594